CLINICAL TRIAL: NCT02927548
Title: Evaluation of the Efficacy and Safety of Advantage® Strips in Women Stress Urinary Incontinence (SUI )
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 15 01 06
Record Dates: First submitted 2016-09-14; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a single-center retrospective study that evaluates the effectiveness and long-term safety of the TVT tape ( advantage Boston Scientific) in the treatment of stress urinary incontinence in women on a population of 500 patients with a mean follow-up of 6 years.

ELIGIBILITY:
Inclusion Criteria:

* patient who received the laying of a strip ADVANTAGE between 1/1/2015 and 1/6/2012

Exclusion Criteria:

* no

Ages: 29 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient of CHU Nîmes
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-01; Primary Completion 2012-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Patient global improvement scale | 6 years
Complications | 6 years
Urinary symptom questionnaire | 6 years